CLINICAL TRIAL: NCT01816126
Title: One-or Two Person Technique and Quality Performance of Colonoscopy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Valduce Hospital (Other)
Responsible Party: Principal Investigator, Arnaldo Amato, Doctor, Valduce Hospital
Other Study IDs: 01-2013
Record Dates: First submitted 2013-03-12; First posted 2013-03-21 (Estimated); Last update posted 2013-03-21 (Estimated); Status verified 2013-03

CONDITIONS: Colonoscopy Techniques

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- one-operator technique
- two-operator technique

SUMMARY:
Colonoscopy can be performed by a one-operator technique with endoscopist personally advancing and withdrawing the scope or by a two-operators technique, with the GI-assistant doing the physical insertion and withdrawal of the scope directed by the endoscopist. Uncontrolled data report that 1 operator technique is associated with a higher adenoma detection rate, although it is also characterized by a lowwer cecal intubation rate and longer intubation time. The aim of present randomized controlled study was to assess whether one technique is better than the other one in terms of colonoscopy quality performances.

ELIGIBILITY:
Inclusion Criteria:

* adult outpatients colonoscopy for screening or surveillance indications

Exclusion Criteria:

* previous colonic surgery
* poor bowel prep
* inability to provide consent

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: colon cancer screening population
Sampling Method: Non-Probability Sample
Dates: Start 2013-02; Primary Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
adenoma detection rate | 4 months

SECONDARY OUTCOMES:
cecal intubation time | 4 months

OTHER OUTCOMES:
tolerability | 4 months
  * pain assessed by nurse (by means a 4 classes 0 to 4 categorical scale)
  * pain judged by patients (by means a 4 classes 0 to 4 categorical scale )

CONTACTS AND LOCATIONS:
Locations (1):
- Valduce Hospital, Como, Italy